CLINICAL TRIAL: NCT02532322
Title: Efficacy of Intravenous Acetaminophen as Analgesic Adjuvant Therapy in Children Undergoing Posterior Fossa Surgery
Brief Title: Efficacy of Acetaminophen in Posterior Fossa Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: not enough patients meeting criteria
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Srijaya K. Reddy, MD, MBA, MD, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00006330
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Arnold-Chiari Malformation; Posterior Fossa Tumors
MeSH Terms: conditions — Arnold-Chiari Malformation; Infratentorial Neoplasms | interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV acetaminophen (Experimental): IV acetaminophen 15 mg/kg (1.5 mL/kg) IV loading dose prior to incision, followed by a 15 mg/kg (1.5 mL/kg) dose given every 6 hours for the first 24 hours after surgery (total of 4 doses postoperatively)
  Interventions: Drug: IV acetaminophen
- normal saline (Placebo Comparator): normal saline (placebo control) 1.5 mL/kg IV loading dose prior to incision, followed by a 1.5 mL/kg dose given every 6 hours for the first 24 hours after surgery (total of 4 doses postoperatively)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: IV acetaminophen — IV acetaminophen 15 mg/kg (1.5 mL/kg) IV loading dose prior to incision, followed by a 15 mg/kg (1.5 mL/kg) dose given every 6 hours for the first 24 hours after surgery (total of 4 doses postoperatively)
  Other Names: Tylenol; APAP
  Arms: IV acetaminophen
Drug: normal saline — normal saline 1.5 mL/kg IV loading dose prior to incision, followed by a 1.5 mL/kg dose given every 6 hours for the first 24 hours after surgery (total of 4 doses postoperatively)
  Other Names: saline placebo; NS 0.9%
  Arms: normal saline

SUMMARY:
Uncontrolled pain after posterior fossa surgery and associated negative side effects of conventional opioid therapy causes significant morbidity and mortality in infants and children. Intravenous (IV) acetaminophen has been shown to be effective in treating mild to moderate pain, and moderate to severe pain in conjunction with adjuvant opioids in children. However, it is unknown if IV acetaminophen is effective as analgesic adjuvant therapy in children undergoing posterior fossa surgery. In this prospective, randomized controlled trial, the investigators aim to determine whether the addition of IV acetaminophen for 24 hours can lead to reduction in postoperative pain and opioid requirement after neurosurgical procedures of the posterior fossa compared with conventional therapy.

DETAILED DESCRIPTION:
The primary goal of this study is to compare the efficacy of IV acetaminophen to placebo in pediatric patients undergoing posterior fossa surgery, with the primary outcome measure being postoperative opioid requirements (morphine equivalent mg/kg). This will be a prospective, randomized, double blind control trial. The patient, research team, surgeon, and anesthesiologist will all be blinded to the patient's treatment group. Patients will receive either IV acetaminophen or equal volume normal saline (placebo) in the perioperative period.

The interventional component of this study involves the intraoperative and postoperative administration of IV acetaminophen. Intraoperative and postoperative data pertaining to adverse events would be collected for safety monitoring purposes.

Enrolled subjects will be randomized to receive either IV acetaminophen or equal volume saline placebo during surgery and for 24 hours postoperatively. According to a computer-generated table of random number assignments, each patient will be randomly assigned to receive one of the following two treatment groups:

Treatment group 1:

IV acetaminophen 15 mg/kg (1.5 mL/kg) IV loading dose prior to incision, followed by a 15 mg/kg (1.5 mL/kg) dose given every 6 hours for the first 24 hours after surgery (total of 4 doses postoperatively). This dosing regimen was chosen based on pharmacokinetic data and recommended dosing guidelines for IV acetaminophen in children 2 to 12 years of age.

Treatment group 2:

Equal volume of normal saline (placebo control) at the same dose and frequency as treatment group 1.

Loading dose volumes and subsequent doses every 6 hours will be determined based on weight of the patient such that they will receive equal volumes of either IV acetaminophen or saline.

Maintenance of anesthesia, including opioid administration, and perioperative management will proceed as per routine care.

POSTOPERATIVE ANALGESIA

At the completion of surgery, the anesthetic agents will be discontinued as per routine care. Per routine care, after tracheal extubation, morphine (0.05 mg/kg/dose) will be administered as needed by the blinded assessor until the patient appears comfortable, defined as the absence of any verbal or behavioral expression of pain. Patients will then be transferred to the intensive care unit (ICU).

Time of entry into the intensive care unit will be recorded. The following assessments will be recorded at time of admission to the ICU:

* vital signs (heart rate, respiratory rate, blood pressure)
* oxygen saturation
* pain score
* sedation score

As part of routine care for postoperative analgesia, patients will receive morphine sulfate at standard doses (0.05 - 0.1 mg/kg/dose every 3 hours as needed for pain). The frequency and dose of morphine will be adjusted according to the patient's pain score, with a goal to maintain a pain score of < 6. In addition, patients will transition to oral opioids as soon as their diet allows.

The following parameters will be used to measure short-term postoperative analgesia and side effects:

* Daily opioid consumption (mg/kg/24h in morphine equivalent using the conversion)
* Pain scores at rest
* Sedation score
* The incidence of post-operative nausea and vomiting (PONV) will be assessed by the need for rescue antiemetics: i.e. ondansetron or promethazine given as needed.
* The incidence and severity of pruritus will be assessed by the need for rescue anti-pruritic: i.e. diphenhydramine or hydroxyzine given as needed for pruritus
* The incidence of pyrexia (defined as core temperature ≥ 38º Celsius). Ketorolac will be administered 0.5 mg/kg q6h prn as needed for pyrexia as per routine care.

Data collection will continue for up to 72 hours postoperatively.

DATA ANALYSIS

Data will be analyzed to determine the decrease in postoperative opioid requirements with or without IV acetaminophen after posterior fossa surgery as the primary outcome. The investigators hypothesize that IV acetaminophen will decrease postoperative opioid requirements, pain and sedation scores, and opioid-induced side effects in children undergoing posterior fossa surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Any child undergoing posterior fossa surgery, including surgery for Chiari Malformation
2. The subject's American Society of Anesthesiologists physical status is 1, 2 or 3
3. Males and females 2 to 12 years old (minorities will be included) - recommended dosing of IV acetaminophen in children is approved for children 2 to 12 years of age
4. Written informed consent from parent/guardian

Exclusion Criteria:

1. Subjects with known or suspected hypersensitivity reaction to acetaminophen
2. Presence or prior history of a known liver disease or coagulation disorder:
3. History of abnormal liver function
4. History of prior liver transplantation
5. Subjects who are on anticoagulant therapy (Coumadin, heparin, aspirin, etc.)
6. History of prior acetaminophen overdose
7. Subjects with the need for mechanical ventilation prior to surgery or postoperatively - unable to assess accurate pain scores in this context
8. The subject has a history or a family (parent or sibling) history of malignant hyperthermia
9. The subject had a recent opioid exposure (within 1 month of surgery)
10. The subject is obese (body mass index >30 kg/m2)
11. The subject is an American Society of Anesthesiologist physical status classification of 4 or greater
12. The subject is scheduled for a surgical sub-procedure
13. Subjects who have been previously enrolled in this protocol may not be enrolled again

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Daily opioid consumption (mg/kg/24 hours using morphine equivalent) | 72 hours postoperatively
  Equianalgesic conversion of opioid consumption to morphine equivalent will be used

SECONDARY OUTCOMES:
Average daily pain scores using Wong-Baker Faces or Numeric Pain Scale | 72 hours postoperatively
  Scores range from 0 [no pain] to 10 [worst possible pain]
Average daily sedation scores using University of Michigan Sedation Scale | 72 hours postoperatively
  Score range from 0 [completely awake] to 4 [asleep but not responsive to any stimuli]
Incidence of opioid-induced side effects | 72 hours postoperatively
  1. Incidence of postoperative nausea and vomiting (PONV) will be assessed by the need for rescue antiemetics (i.e. ondansetron or promethazine given as needed)
  2. Incidence and severity of pruritus will be assessed by the need for rescue anti-pruritic (i.e. diphenhydramine or hydroxyzine given as needed for pruritus)

CONTACTS AND LOCATIONS:
Overall Officials: Srijaya K Reddy, MD, MBA, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Benedittis G, Lorenzetti A, Migliore M, Spagnoli D, Tiberio F, Villani RM. Postoperative pain in neurosurgery: a pilot study in brain surgery. Neurosurgery. 1996 Mar;38(3):466-9; discussion 469-70. doi: 10.1097/00006123-199603000-00008. PMID 8837797
- [Background] Morad A, Winters B, Stevens R, White E, Weingart J, Yaster M, Gottschalk A. The efficacy of intravenous patient-controlled analgesia after intracranial surgery of the posterior fossa: a prospective, randomized controlled trial. Anesth Analg. 2012 Feb;114(2):416-23. doi: 10.1213/ANE.0b013e31823f0c5a. Epub 2011 Dec 9. PMID 22156333
- [Background] Baley K, Michalov K, Kossick MA, McDowell M. Intravenous acetaminophen and intravenous ketorolac for management of pediatric surgical pain: a literature review. AANA J. 2014 Feb;82(1):53-64. PMID 24654353
- [Background] Alhashemi JA, Daghistani MF. Effect of intraoperative intravenous acetaminophen vs. intramuscular meperidine on pain and discharge time after paediatric dental restoration. Eur J Anaesthesiol. 2007 Feb;24(2):128-33. doi: 10.1017/S0265021506001232. Epub 2006 Aug 8. PMID 16895621
- [Background] Alhashemi JA, Daghistani MF. Effects of intraoperative i.v. acetaminophen vs i.m. meperidine on post-tonsillectomy pain in children. Br J Anaesth. 2006 Jun;96(6):790-5. doi: 10.1093/bja/ael084. Epub 2006 Apr 13. PMID 16613928
- [Background] Lahtinen P, Kokki H, Hendolin H, Hakala T, Hynynen M. Propacetamol as adjunctive treatment for postoperative pain after cardiac surgery. Anesth Analg. 2002 Oct;95(4):813-9, table of contents. doi: 10.1097/00000539-200210000-00005. PMID 12351250